CLINICAL TRIAL: NCT04126174
Title: Femtosecond Laser-assisted Arcuate Incisions Versus Manual Arcuate Incisions Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gainesville Eye Associates (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB-19-001
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-02

CONDITIONS: Cataract
Keywords: astigmatism, limbal relaxing incisions
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Intervention Model Description: Contralateral eye study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Femtosecond limbal relaxing incision (LRI) (Active Comparator): Eyes will be treated with arcuate incisions from a femtosecond laser system.
  Interventions: Device: femtosecond laser system arcuate corneal incision
- Manual LRI (Active Comparator): Eyes will be treated with arcuate incisions completed manually with a blade.
  Interventions: Other: Manual LRI

INTERVENTIONS:
Device: femtosecond laser system arcuate corneal incision — Corneal arcuate incision made either with a blade (manual) or femtosecond laser system.
  Other Names: LRI
  Arms: Femtosecond limbal relaxing incision (LRI)
Other: Manual LRI — Manual LRI
  Arms: Manual LRI

SUMMARY:
This study is designed to compare the effectiveness of LenSx laser arcuate relaxing incisions vs. manual (blade) arcuate relaxing incisions in patients with low, but significant, levels of astigmatism.

DETAILED DESCRIPTION:
This study is a comparative, prospective, randomized contralateral eye study of visual outcomes after LenSx laser arcuate relaxing incisions utilizing the Woodcock nomogram at 90% thickness vs. manual (blade) fixed keratome diamond knife at 600 microns for arcuate relaxing incisions utilizing the Donnenfeld nomogram. Subjects will be assessed pre-operatively and at 1 day, 1 month and 3 months post-operatively. Clinical evaluations will include measurement of visual acuity, manifest refraction and corneal astigmatism measurement with the Lenstar and slit lamp exam.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* are willing and able to understand and sign an informed consent;
* are willing and able to attend all study visits;
* are more than 40 years of age, of either gender and any race;
* are presenting for cataract surgery or refractive lens exchange with a desire to reduce astigmatism and will be implanted with a non-toric lens
* have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract)
* have 0.50 D to 1.75 D of regular corneal astigmatism
* have potential acuity of 20/25 or better
* Are scheduled to have a non-toric monofocal intraocular lens (IOL) (SN60WF) lens implanted in both eyes

Exclusion Criteria If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Irregular astigmatism (e.g. keratoconus)
* Corneal pathology (e.g. scar, dystrophy, pterygium, moderate-to-severe dry eye)
* Monocular status (e.g. amblyopia)
* Previous radial keratotomy, corneal refractive surgery or other corneal surgery (e.g. corneal transplant, lamellar keratoplasty)
* Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy)
* Diabetic retinopathy
* Macular pathology (e.g. age-related macular degeneration, epiretinal membrane)
* History of retinal detachment
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect post-operative visual acuity.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton G Blehm, MD, Principal Investigator — Gainesville Eye Associates
Locations (1):
- Gainesville Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eye
Groups:
- Femtosecond Limbal Relaxing Incision (LRI): Eyes will be treated with arcuate incisions from a femtosecond laser system.
  femtosecond laser system arcuate corneal incision: Corneal arcuate incision made with a femtosecond laser system.
Period: Overall Study
Arm/Group | Femtosecond Limbal Relaxing Incision (LRI) | Manual LRI
Started | 41; 41 Eye | 41; 41 Eye
Completed | 38; 38 Eye | 38; 38 Eye
Not Completed | 3; 3 Eye | 3; 3 Eye
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Only subjects who completed the study are included in the baseline analysis.
Groups:
- All Participants: Corneal arcuate incision made either with a blade (manual) or femtosecond laser system.
Arm/Group | All Participants
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only subjects completing the study were included in the baseline analysis.
  years | 69 (7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only subjects completing the study were included in the baseline analysis.
  Participants
    Female | 21
    Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: Only subjects completing the study were included in the analysis population.
  Participants
    United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Residual Refractive Astigmatism
Description: Residual refractive astigmatism measured in diopters
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Femtosecond Limbal Relaxing Incision (LRI) | Manual LRI
Number analyzed (Participants) | 38 | 38
Number analyzed (Eyes) | 38 | 38
diopters | .21 (.33) | .22 (.31)

2. Secondary Outcome: Eyes With Residual Refractive Astigmatism < 0.50 Diopters (D)
Description: The number of eyes with residual refractive astigmatism < 0.50 diopters (D)
Time Frame: 3 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Femtosecond Limbal Relaxing Incision (LRI) | Manual LRI
Number analyzed (Participants) | 38 | 38
Number analyzed (Eyes) | 38 | 38
Eyes | 36 | 34

3. Secondary Outcome: Uncorrected Monocular Distance Visual Acuity
Description: Uncorrected monocular distance visual acuity in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Femtosecond Limbal Relaxing Incision (LRI) | Manual LRI
Number analyzed (Participants) | 38 | 38
Number analyzed (Eyes) | 38 | 38
logMAR | .1 (.12) | .08 (.10)

4. Secondary Outcome: Spherical Equivalent Refraction
Description: Spherical equivalent refraction in diopters
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Femtosecond Limbal Relaxing Incision (LRI) | Manual LRI
Number analyzed (Participants) | 38 | 38
Number analyzed (Eyes) | 38 | 38
diopters | -.02 (.37) | 0 (.27)

5. Secondary Outcome: Corneal Astigmatism
Description: Anterior corneal astigmatism
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Femtosecond Limbal Relaxing Incision (LRI) | Manual LRI
Number analyzed (Participants) | 38 | 38
Number analyzed (Eyes) | 38 | 38
diopters | .63 (.34) | .7 (.4)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Femtosecond Limbal Relaxing Incision (LRI) | Manual LRI
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 2/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Femtosecond Limbal Relaxing Incision (LRI) (N=41) | Manual LRI (N=41)
Full thickness perforation (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT04126174/Prot_SAP_000.pdf